CLINICAL TRIAL: NCT04875104
Title: A Randomized Clinical Trial on Upper Sequential Distalization With Temporary Anchorage Devices (TADs) and Two Aligner Systems
Brief Title: Upper Sequential Distalization With TADs and Aligners
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URI 39-150221
Record Dates: First submitted 2021-04-21; First posted 2021-05-06 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-04

CONDITIONS: Malocclusion, Angle Class II; Distalization
Keywords: Dentistry; Orthodontics; Clear aligner therapy; Aligners; Invisalign; Upper molar distalization; Temporary anchorage devices; Mini-screws
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — Orthodontics

STUDY DESIGN:
Intervention Model Description: This study will be a 4-arm parallel-group, randomized, prospective superiority clinical trial with an allocation ratio of 1:1:1:1 There will be four groups of aligners of different brands.
Masking Description: Patients recruited into the study who met the inclusion criteria will be assigned to group 1 Invisalign, group 2 Spark, group 3 Quicksmile or group 4 ClearCorrect. To generate the allocation sequence, a block randomization system with block sizes of 4 and a 1:1:1:1 allocation ratio will be applied using GraphPad online software. The allocation will be concealed from the orthodontist, investigator, and patient. When a patient was determined to be eligible, the orthodontist explained the clinical trial to them, and the patient signed the informed consent to participate. After the allocation of the interventions, neither the patient nor the orthodontist will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Invisalign (Active Comparator): Patients treated with Invisalign aligners
  Interventions: Device: Orthodontic treatment with Invisalign system
- Spark (Experimental): Patients treated with Spark aligners
  Interventions: Device: Orthodontic treatment with Spark system
- Quicksmile (Experimental): Patients treated with Quicksmile aligners
  Interventions: Device: Orthodontic treatment with Quicksmile system
- ClearCorrect (Experimental): Patients treated with ClearCorrect aligners
  Interventions: Device: Orthodontic treatment with ClearCorrect system

INTERVENTIONS:
Device: Orthodontic treatment with Invisalign system — Patients are going to receive an orthodontic treatment with Invisalign aligners.
  Arms: Invisalign
Device: Orthodontic treatment with Spark system — Patients are going to receive an orthodontic treatment with Spark aligners.
  Arms: Spark
Device: Orthodontic treatment with Quicksmile system — Patients are going to receive an orthodontic treatment with Quicksmile aligners.
  Arms: Quicksmile
Device: Orthodontic treatment with ClearCorrect system — Patients are going to receive an orthodontic treatment with ClearCorrect aligners.
  Arms: ClearCorrect

SUMMARY:
In this study the investigators are going to compare the predictability of the backward movement of upper first molars in patients with the upper dentition more advanced than the lower dentition. The investigators are going to study if the movements that they predict are achieved and in which proportion and compare it between four different aligner systems. The investigators hypothesis is that there are no differences in the predictability of this movement between the four aligner systems.

DETAILED DESCRIPTION:
In this study the investigators are going to assess and compare the predictability of distal movement of upper molars in patients with class II molar relationship when superimposing the initial malocclusion with the real end of distalization phase and the predicted end of distalization phase. Also, the investigators are going to study another dental movements, pain level, aligner properties, oral hygiene, posterior root resorption, patient satisfaction, quality of life and efficiency of these systems.

The aligner systems that are going to be used are Invisalign System (Align Technology, San José, CA), Spark Aligners (Ormco, Glendora, CA), Quicksmile (Madrid, España) and ClearCorrect (Straumann, Austin, TX). To help achieve the molar movement there is going to be place a TAD (temporary anchorage device) between two teeth. Before starting the study, the patients will need some pretreatment records (radiographs, photographs, dental casts and intraoral scan) to make a diagnosis and confirm if the patient is suitable for the study.

The required sample will be 98 subjects, assuming a sample loss of 15% the required sample will be 115 subjects per group. Patients will be randomly assigned to either group using a block randomization system and carried out by a researcher not involved in the study. Data normality will be examined with the Kolmogorov-Smirnov. Descriptive statistics of the different outcomes will be calculated for each group. Student's paired sample t-test will be used to analyze intragroup differences between T0 and T1. Intergroup comparison among different intervention groups will be performed using multiple analysis of variance (MANOVA), with Tukey's post-hoc test. The investigators will use the Pearson correlation coefficient to evaluate the linear relationship between the mm of distalization achieved and the mm of crowding and between the mm of distalization achieved and the patients age. The investigators will perform a binary logistic regression in order to assess the influence of confounding factor (clinical variables) on the primary outcome. All statistical analysis will be conducted using IBM SPSS 24.0 (SPSS Inc., Chicago, IL, USA) software with a 0.05 level of significance.

ELIGIBILITY:
Inclusion Criteria:

* Patients who needed orthodontic treatment with aligners in both jaws.
* Adult patients (>18 years)
* Full permanent dentition (excluding third molars)
* Patients with non-surgical or non-extraction (excluding third molars) treatment
* No active periodontal disease
* Patients with class II molar relationship that needed molar distalization

Exclusion Criteria:

* Patients with systemic diseases affecting bone metabolism or teeth or inflammatory diseases
* Patients undergoing treatment with immunosuppressant or bisphosphonates
* Patients undergoing chemo and radiotherapy
* Patients with any other syndrome-associated orofacial deformation, cleft lip or palate
* Pregnant women or non(or poor)-compliance patients with skeletal discrepancies
* Patients with dental or skeletal crossbite that need 3 mm or more per side of expansion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Predictability of upper molar distalization | Time 0 (initial day of treatment) to Time 1 (achievement of class I, 10-12 months)
  Predictability of upper molar distalization will be assessed in mm comparing pre- and post-distalization 3D models. Pre-treatment 3D model (ModT0) will be superimposed with ideal end of distalization model (ClinT1) and real end of distalization models to see how much distalization has been achieved. The predictability will be the difference between the achieved and the expected amount of tooth movement and to quantify distalization measurements are going to be made in various views and teeth.
Achievement of molar class I | Time 0 (initial day of treatment) to Time 1 (achievement of class I, 10-12 months)
  Achievement of class I after distalization will be assessed with yes (=1) or no (=0). It will be considered class I when the mesiobuccal cusp of the upper first molar occludes with the mesiobuccal groove of the lower first molar when seeing models in occlusion with a discrepancy of 0.5 mm.

SECONDARY OUTCOMES:
Individual tooth movement | Time 0 (initial day of treatment) to Time 1 (achievement of class I, 10-12 months)
  Individual tooth movement will be evaluated comparing pre- and post distalization 3D models. In the same superposition procedure explained in the previous section, we are going to study the individual movements of the teeth to see where and which movements have not been achieved. And, the difference between the achieved and the expected amount of tooth movement was calculated. We will quantify the accuracy of each individual movement and we will obtain an index of the accuracy of each movement and the movement will be more precise when the value is closer to 1.
Periodontal mucosa health status - Plaque Index (PI) | Time 0 (initial day of treatment), month 3 and month 6
  Periodontal health status measurements will be made on the right maxillary first molar, premolar and central incisor before treatment and after one, three and six months during treatment in both aligner systems. To assess plaque index (PI) the accumulation of plaque will be visually inspected in the gingival area and will be classified on a score of 0 to 3 of the modified index of Löe, where 0 will be "no plaque on inspection/probing" and 3 will be "presence of a thick layer of plaque".
Periodontal mucosa health status - Gingival Index (GI) | Time 0 (initial day of treatment), month 3 and month 6
  Periodontal health status measurements will be made on the right maxillary first molar, premolar and central incisor before treatment and after one, three and six months during treatment in both aligner systems. Color and tissue consistency will be evaluated according to the severity of the inflammation of the gingival margin and will be classified on a score of 0 to 3 of the modified index of Löe, were 0 is "Physiologic gingiva" and 3 is "severe inflammation".
Periodontal mucosa health status - Papillary Bleeding Index (PBI) | Time 0 (initial day of treatment), month 3 and month 6
  Periodontal health status measurements will be made on the right maxillary first molar, premolar and central incisor before treatment and after one, three and six months during treatment in both aligner systems. The PBI will be assessed by inserting a periodontal probe into the gingival sulcus of those three teeth and waiting 20 seconds after probing and will be classified on a score of 0 to 3 of the modified index of Löe, were 0 is "no bleeding" and 3 is "profuse bleeding".
Peri-implant mucosa inflammation | Time 0 (initial day of treatment), month 3 and month 6
  Peri-implant mucosa health status will be also assessed as a reaction of pressure around the TAD with a periodontal probe and registering bleeding with Absence=0 or Presence=1.
TADs stability | Time 0 (initial day of treatment), month 3 and month 6
  Stability will be evaluated in each appointment with cotton tweezers and there will be two groups: mobile (yes=1) and not mobile (no=1). TAD failure will be considered when the implant loosened before or during completion of its use, when it presents mobility or pain on percussion.
Quantification of the modulus of elasticity | Time 0 (initial day of treatment) and week 2
  Modulus of elasticity measures resistance to being deformed elastically when a stress is applied to it. This will be evaluated on samples cut out from as-received aligners and on aligners after two weeks of use with instrumented indentation testing using a universal testing machine.
Quantification of changes in force after 75 desinsertion cycles | Time 0 (initial day of treatment) and week 2
  The desinsertion force is the force that it is necessary to remove the aligners from de teeth (N). This will be evaluated in vitro in the first passive aligner after being subjected to 75 cycles of insertion/desinsertion of its stereolithographic using a universal testing machine.
Quantification of changes in desinsertion time after 75 desinsertion cycles | Time 0 (initial day of treatment) and week 2
  The desinsertion time is the time that it is necessary to remove the aligners from de teeth (s). This will be evaluated in vitro in the first passive aligner after being subjected to 75 cycles of insertion/desinsertion of its stereolithographic using a universal testing machine.
Quantification of changes in deformation after 75 desinsertion cycles | Time 0 (initial day of treatment) and week 2
  The deformation of the aligner is the amount of deformation that an aligner undergoes when it is removed (mm). This will be evaluated in vitro in the first passive aligner after being subjected to 75 cycles of insertion/desinsertion of its stereolithographic using a universal testing machine.
Quantification of the aligner fit on the attachments | Time 0 (initial day of treatment) and week 2
  The aligner fit is the distance between the internal surface of the aligner and the teeth or attachments. This is use to study the gap between the aligners and the teeth. This will be evaluated in vitro in the passives aligners as-received and after being subjected to 75 cycles of insertion/desinsertion of its stereolithographic using a universal testing machine.
Orthodontically induced external apical root resorption (OIEARR) | Time 0 (initial day of treatment) and month 6
  OIEARR will be measured on upper posterior teeth root lengths before and after distalization with the use of panoramic radiographs. They were divided into two groups (presence>2mm/absence<2mm).
Quantification of pain level | Week 3, week 7 and week 11.
  Pain level will be assessed using a 0-10 numerical pain rating scale where 0 is "no pain" and 10 is "worst possible pain". They will also be asked some questions regarding pain evaluation and finally, their analgesic consumption, type and frequency. They have to be completed each day during the third week, in week 7 and 11.
Quantification of quality of life (OHIP-14sp) | Time 0 (initial day of treatment) and month 1
  Quality of life will be evaluated with the Spanish version of the Oral Health Impact Profile-14 (OHIP-14sp). It is a 14 item questionnaire in which participants have to respond a 5-point Likert scale coded for: never (0), hardly ever (1), occasionally (2), fairly often (3) and very often (4). The overall OHIP-14sp outcome will be obtained by summing the items and so the score ranges from 0 to 56 and the higher the score the higher the lever of oral quality of life and vice versa.
Quantification of patient satisfaction (DSQ) | Time 0 (initial day of treatment) and month 1
  Dental Satisfaction Questionnaire (DSQ) will be used to study patient satisfaction. It has 19 items with a Likert scale from 1 to 5, were 1 is "agree completely", 2 "agree", 3 "undecided", 4 "disagree" and 5 "disagree completely". Agree completely responses were rated with 5 points and disagree completely with 1. The overall outcome will be obtained by summing the items and so the score ranges from 19 to 95, having into account that items 1, 3, 4, 5, 8, 11, 13 and 17 are reverse scored. The higher the score the higher the level of patient satisfaction and vice versa.
Quantification of the treatment and chair time. | Time 0 (initial day of treatment) to Time 1 (achievement of class I, 10-12 months)
  Distalization treatment time will be measured in months and days since the first aligner is delivered to the patient until the last day of distalization of the first premolar. It should be taken into consideration the mid-course corrections if necessary.
  Chair time of each scheduled or non-scheduled appointment is the total time that the patient spends in the dental chair regardless of the interaction with the doctor or assistant. Treatment time in minutes will be estimated with a stopwatch and rounded up to the nearest 30 seconds.
Quantification of the number of appointments. | Time 0 (initial day of treatment) to Time 1 (achievement of class I, 10-12 months)
  Total number of appointments, emergency visits related to the appliances and cancellations will be also noted. Regarding the emergency visits the reason will be noted, attachment debonding, damage or loss of the aligners or other reasons related with the TADs.
Quantification of the direct and indirect costs. | Time 0 (initial day of treatment) to Time 1 (achievement of class I, 10-12 months)
  Direct costs (Euros) in this study included material costs and treatment time needed. Indirect costs (Euros) will be defined as loss of income, assuming that the patients will be absent from work during the orthodontic appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Iglesias Linares, Study Director — Universidad Complutense de Madrid
Locations (1):
- Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
We have not yet decided the format in which to share the information.